CLINICAL TRIAL: NCT07393685
Title: Effect of Xuanfei Jiangzhuo Decoction on Clinical Remission in Influenza-Induced AECOPD: Study Protocol for a Prospective, Real-World Cohort Study
Brief Title: Effectiveness of Xuanfei Jiangzhuo Decoction for Influenza-Induced AECOPD: A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Yanqi Song, Ph.D, Tianjin Medical University
Other Study IDs: IRB2025-YX-643-01; IRB2025-YX-643-01 (Other Grant/Funding Number: Tianjin Medical University General Hospital)
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Influenza, Human; Virus Diseases
Keywords: COPD Exacerbation; Real-World Study; Traditional Chinese Medicine
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — yifei xuanfei jiangzhuo; Oseltamivir; baloxavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure Group: XFJZD + Western Medicine: Patients diagnosed with influenza-induced AECOPD who choose to receive Xuanfei Jiangzhuo Decoction (XFJZD) combined with standard Western medicine based on personal preference and physician recommendations. XFJZD is administered orally as a liquid decoction, 200 mL per dose, twice daily for 5 days. They also receive standard antiviral therapy (Oseltamivir or Baloxavir marboxil) and routine COPD maintenance therapy.
  Interventions: Drug: Xuanfei Jiangzhuo Decoction; Drug: Standard Antiviral Therapy (Oseltamivir or Baloxavir marboxil)
- Non-Exposure Group: Standard Western Medicine: Patients diagnosed with influenza-induced AECOPD who choose to receive standard Western medicine alone based on personal preference. This includes standard antiviral therapy (Oseltamivir or Baloxavir marboxil) and routine maintenance therapy for COPD (e.g., ICS/LABA/LAMA, theophylline, roflumilast). This group does not receive the XFJZD intervention.
  Interventions: Drug: Standard Antiviral Therapy (Oseltamivir or Baloxavir marboxil)

INTERVENTIONS:
Drug: Xuanfei Jiangzhuo Decoction — A traditional Chinese medicine composite formula derived from Maxing Shigan Tang and Shengjiang San. It is administered orally as a liquid decoction, 200 mL per dose, twice daily (morning and evening, 30 minutes after meals) for 5 days.
  Groups: Exposure Group: XFJZD + Western Medicine
Drug: Standard Antiviral Therapy (Oseltamivir or Baloxavir marboxil) — Patients receive standard antiviral treatment according to clinical guidelines and physician judgment. Medications include Oseltamivir (e.g., 75 mg twice daily for 5 days) or Baloxavir marboxil (singl

SUMMARY:
The goal of this observational study is to learn if a traditional Chinese herbal medicine (Xuanfei Jiangzhuo Decoction) works to help older adults recover from a COPD flare-up caused by the flu (influenza virus). The main questions it aims to answer are:

Does the herbal medicine help participants feel better and recover faster? Does it lower the chance of getting a second infection from bacteria? Is the herbal medicine safe to use? Researchers will compare participants who choose to take the herbal medicine along with their standard flu treatment (Oseltamivir or Baloxavir) to participants who only take the standard flu treatment (Oseltamivir or Baloxavir).

Participants will:

Take the herbal medicine (a liquid drink) twice a day for 5 days, or just take their standard flu medicine for 5 days.

Visit the clinic 4 times over 28 days for checkups and tests. Provide blood and stool samples to help researchers understand how the medicine affects the body and gut health.

Answer simple questions about their cough, breathing, and energy levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD and currently in an acute exacerbation phase according to the Guidelines for the Diagnosis and Treatment of COPD (2021 Revision).
* Confirmed influenza virus infection (Type A or B) via rapid antigen test or PCR within 48 hours of onset.
* Aged 60 years or older.
* Voluntarily participate and provide written informed consent.
* Eligible for pharmacotherapy (able to take TCM combined with Western medicine or Western medicine alone).

Exclusion Criteria:

* Known allergy or hypersensitivity to any component of the study medications (XFJZD or standard Western antiviral agents).
* Presence of severe bacterial co-infection at enrollment requiring systemic antibiotic therapy.
* Severe dysfunction of major organs that may interfere with efficacy or safety assessment (e.g., severe cardiac insufficiency, hepatic impairment, or renal failure).
* Participation in other interventional clinical trials within the past 3 months.
* Inability to be contacted for follow-up (e.g., lack of permanent address or valid contact information).
* Any other condition that, in the opinion of the investigator, would make the patient unsuitable for study participation (e.g., severe cognitive impairment or psychiatric disorders).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years or older presenting with influenza-induced Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD) at the Department of Traditional Chinese Medicine and the Department of Infectious Diseases at Tianjin Medical University General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Remission of AECOPD | From baseline (Day 0) up to Day 28
  Defined as the duration from treatment initiation to the point where the modified Medical Research Council (mMRC) dyspnea scale score returns to the patient's pre-exacerbation baseline, and major respiratory symptoms (cough and dyspnea) show stable improvement for at least 48 hours. The mMRC scale ranges from 0 to 4, with higher scores indicating more severe breathlessness.

SECONDARY OUTCOMES:
Time to Defervescence | From baseline (Day 0) up to Day 14
  Defined as the time until axillary temperature is ≤ 37.4°C and maintained for 24 hours.
Time to Alleviation of Individual Symptoms | From baseline (Day 0) up to Day 28
  Defined as the time until individual symptom scores are ≤ 1 and maintained for 24 hours.
Change in COPD Assessment Test (CAT) Score | Baseline (Day 0), Day 5, Day 14, and Day 28
  The CAT measures the impact of COPD on a person's life. Scores range from 0-40, with higher scores indicating a more severe impact of the disease.
Rate of Secondary Bacterial Infection | From baseline (Day 0) through Day 28
  Percentage of participants with confirmed secondary bacterial infection verified by blood routine, sputum culture, or blood culture.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided